CLINICAL TRIAL: NCT03421184
Title: Dietary Phytoestrogens in Blood and Urine of Female Patient With Acute Systemic Lupus Erythematosus
Brief Title: Dietary Phytoestrogens as Risk Factors for Systemic Lupus Erythematosus
Acronym: ISOLED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2017/18
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Lupus Erythematosus; Rheumatoid Arthritis; Autoimmune Thrombocytopenia
Keywords: autoimmune disease; endocrine disruptors; isoflavones; lignans; diet exposure; risk factor
MeSH Terms: conditions — Arthritis, Rheumatoid; Purpura, Thrombocytopenic, Idiopathic; Autoimmune Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patient with Systemic Lupus Erythematosus (Experimental): 30 women with SLE
  Interventions: Other: blood sample; Other: urine sample; Other: food questionnaire; Other: hair
- Patients with other autoimmune diseases (Active Comparator): 20 patients with rheumatoid arthritis, 20 patients with autoimmune thrombocytopenia
  Interventions: Other: blood sample; Other: urine sample; Other: food questionnaire; Other: hair
- Healthy control (Active Comparator): 30 healthy control women
  Interventions: Other: blood sample; Other: urine sample; Other: food questionnaire; Other: hair

INTERVENTIONS:
Other: blood sample — 25 ml whole blood for Peripheral blood mononuclear cell (PBMC) and monocytes isolation
Other: urine sample — 10 ml
Other: food questionnaire — dietary habit enquiry and a 48h dietary
Other: hair — lock of hair

SUMMARY:
The study aims at determining if dietary phytoestrogens can be risk factors for Systemic Lupus Erythematosus (SLE). Dietary enquiry and phytoestrogens measurements will be performed in blood and urine of patients with SLE in an active phase of the disease, in patient with other autoimmune diseases and in healthy volunteers. Subjects will be premenopausal women and when possible at a define stage of the menstrual cycle. Free blood estradiol will be assayed as a confounding risk factor.

DETAILED DESCRIPTION:
SLE is a disease occurring in 90% of the cases in pre-menopausal women. The causing factors are largely unknown even though genetic and environmental factors have already been identified. Estrogens, on one side, have been shown to negatively influence the incidence and severity of the disease while testosterone and progesterone on the other side are thought to be protective. Endocrine disruptors can potentially influence the occurrence and severity of the disease. Among these disruptors, soy isoflavones which are ubiquitous in modern processed food are known to be estrogenic and anti-androgenic. Their depleting effect on luteinizing hormone (LH) secretion can also lead to progesterone plasma level impairments. For these reasons, estrogenic isoflavones, appear as potential environmental risk factors for SLE and its flares. Although some data exist in transgenic rodent, there is actually no clinical data in young women.

The study is an observational, monocentric, preliminary study aiming at determining if estrogenic isoflavones can be risk factors for SLE. No treatment is planned. The intervention will be the collection of extra blood and urine samples on SLE subjects and on autoimmune and healthy counterparts.

Consumers are unintentionally exposed to estrogenic isoflavones through their diet. A dietary habit enquiry and a 48h dietary recall (based on pharmacokinetics of soy-isoflavones) will be proposed to the included subjects. Urine and blood samples collected during a clinical visit performed 7 days after the onset of previous menses will be analyzed for soy isoflavones, metabolites and for enterolactone both free and conjugated. Free estradiol will be assayed as a potential confounding risk factor.

ELIGIBILITY:
Inclusion Criteria:

* Group : Systemic Lupus Erythematosus :

  * Premenopausal women over 18
  * with acute LEAD flare
  * having given informed consent
  * and being covered by social insurance.
* Group : Autoimmune diseases :

  * Premenopausal women of matching age with other autoimmune disease,
  * having given informed consent
  * and being covered by social insurance.
* Healthy controls :

  * Premenopausal women over 18,
  * having given informed consent,
  * and being covered by social insurance.

Exclusion Criteria:

* Group Systemic Lupus Erythematosus and group autoimmune diseases

  * Human Immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis C virus (HBV) sero-positivity;
  * pregnant or lactating women;
  * menopausal women;
  * patient in remission of quiescent phase of her pathology;
* Healthy controls :

  * HIV, HCV or HBV sero-positivity;
  * pregnant or lactating women;
  * menopausal women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Quantification of different isoflavones and enterolactone | At baseline (day 0)
  in the blood and urine of patients and healthy controls

SECONDARY OUTCOMES:
Quantification of free estradiol concentrations | At baseline (day 0)
  in the blood and urine of patients and healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François VIALLARD, Prof, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - service de médecine interne, Pessac, France